CLINICAL TRIAL: NCT02085252
Title: An Open-Label, Multicenter, Phase III Study to Assess the Impact of Transient Androgenic Deprivation With Enantone LP 11.25 Mg (Leuprorelin) on the Histological Progression of Indolent Prostate Cancer
Brief Title: A Study of the Effect of Enantone LP 11.25 mg (Leuprorelin) on the Histological Progression of Indolent Prostate Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FR-LEU-002; 2012-002653-35 (EudraCT Number); U1111-1146-5402 (Registry Identifier: WHO)
Record Dates: First submitted 2013-07-24; First posted 2014-03-12 (Estimated); Results first posted 2019-04-16 (Actual); Last update posted 2019-06-28 (Actual); Status verified 2019-06

CONDITIONS: Prostate Cancer
Keywords: Drug Therapy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Leuprolide; bicalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Leuprorelin 11.25 mg (Experimental): Active surveillance after a single subcutaneous injection of leuprorelin 11.25 mg and bicalutamide 50 mg, tablet, orally, once daily, to prevent flare-up for 15 days.
  Interventions: Drug: Leuprorelin; Drug: Bicalutamide
- Active surveillance (No Intervention): Active surveillance is close medical monitoring of prostate cancer for any changes.

INTERVENTIONS:
Drug: Leuprorelin — Solution for injection
  Other Names: Enantone ®
  Arms: Leuprorelin 11.25 mg
Drug: Bicalutamide — Bicalutamide tablets
  Other Names: Casodex ®
  Arms: Leuprorelin 11.25 mg

SUMMARY:
The purpose of this study is to assess two treatment strategies (leuprorelin treatment and active surveillance without androgen deprivation) for indolent prostate cancer and to compare their therapeutic benefit for management of patients with low-risk, localized prostate cancer.

DETAILED DESCRIPTION:
The drug being tested in this study is called leuprorelin. Leuprorelin is being tested to treat people who have prostate cancer. Study assessments will include adverse events, prostatic-specific antigen (PSA) levels, and prostate biopsies.

The study will enroll approximately 120 patients. Participants will be randomly assigned (by chance, like flipping a coin) to a treatment group that will receive leuprorelin 11.25 mg (as one injection) or to an untreated observation group. Patients in the leuprorelin group will also receive bicalutamide 50 mg, a non-steroidal antiandrogen, once daily for 15 days to prevent a flare-up.

This multi-center trial will be conducted in France. The overall time to participate in this study is 12 months. After the screening visit, participants will make 6 visits to the clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Is an out-patient 50 to 80 years old.
2. Has read, understood, signed and dated the informed consent.
3. Has indolent prostate cancer defined by:

   * Clinical Stage T1c or T2a.
   * Biopsy cores of which at least 12 reveal the presence of positive cores and the absence of cores with tumor length > 3 mm.
   * Absence of Grade 4 cells (Gleason <7).
   * Prostate specific antigen (PSA) levels <10 ng/ml.
4. Has a life expectancy > 5 years.
5. Has accepted the principle of active surveillance.
6. Is willing to participate in the study for a minimum of fifteen months.

Exclusion Criteria:

1. Has prior androgen deprivation including a 5-alpha reductase inhibitor (finasteride or dutasteride) within the last 6 months.
2. Has psychological failure related to prostate cancer therapy.
3. Has any active disorder likely to affect the conduct of the study or the patient's prognosis during the study.
4. Has a mental deficiency or any other reason that may hinder the understanding or strict application of the protocol.
5. Is under judicial protection, tutorship or curatorship.
6. Is unlikely to attend control visits.
7. Is currently enrolled in an investigational study or has participated in another investigational study within the last 3 months.
8. Has an allergy or hypersensitivity to any components of leuprorelin (Enantone LP) 11.25 mg or Casodex® 50 mg.
9. Has a medical history of severely impaired hepatic function linked to bicalutamide or a pathological cause.
10. Has testosterone level < 0.5 ng/ml.

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2013-06-03 (Actual); Primary Completion 2016-11-08 (Actual); Study Completion 2016-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (2):
- France (2):
  - Tenon Hospital Paris France, Paris
  - Ouzid, Paris La Défense,, Paris

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 22 investigative sites in France from 03 June 2013 to 08 November 2016.
Pre-assignment Details: Participants with a diagnosis of Prostate Cancer were randomised equally to one of two arms: leuprorelin 11.25 mg or active surveillance. 116 participants were randomized but 1 patient was excluded due to absence of prostate cancer before treatment.
Period: Overall Study
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance
Started | 58 | 57
Completed | 57 | 53
Not Completed | 1 | 4
Not completed — Withdrawal of Consent | 1 | 0
Not completed — Adverse Event | 0 | 1
Not completed — Discontinuation Due to Patient Decision | 0 | 1
Not completed — Reason Not Specified | 0 | 1
Not completed — Reason Unknown | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full Analysis Set included all participants with prostate cancer who signed informed consent and were randomised.
Groups:
- Total: Total of all reporting groups
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance | Total
Number analyzed (Participants) | 58 | 57 | 115
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.22 (5.76) | 63.60 (5.56) | 64.92 (5.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 58 | 57 | 115
Region of Enrollment [Count of Participants; unit: Participants]
  France | 58 | 57 | 115
Height [Mean (Standard Deviation); unit: centimeters (cm)] — Population: Number analyzed is the number of participants with data available for analysis for this baseline measure.
  centimeters (cm)
    number analyzed (Participants) | 54 | 54 | 108
    (all) | 171.85 (6.55) | 173.69 (8.08) | 172.77 (7.38)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Negative Biopsies at Month 12
Description: Staging biopsy of at least 12 cores were sampled and analyzed according to a centralized biopsy procedure which confirm the results of the first biopsy [presence of positive cores, the absence of core with tumor length > 3 millimeters (mm), and absence Grade 4 cells (Gleason score < 7)]. The Gleason score grades prostate cancer tissue, based on its appearance under a microscope. Scores range from 2 to 10, with a higher score meaning that the cancer tissue is more likely to spread.
Time Frame: Month 12
Population: Full Analysis Set included all participants with prostate cancer who signed informed consent and were randomised. Participants with missing biopsy results have been excluded from the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance
Number analyzed (Participants) | 53 | 54
Participants | 28 | 17
Statistical Analysis 1: Comparison: Leuprorelin 11.25 mg vs Active Surveillance; The null hypothesis was that there was no difference between the two treatment strategies; Test type: Superiority or Other; p = 0.0318, Chi-squared — A 2-sided significance level of 5% was used. There was no adjustment for multiple comparisons

2. Secondary Outcome: Number of Participants With Gleason Score ≥ 7
Description: Gleason score grades prostate cancer tissue, based on its appearance under a microscope. Scores range from 2 to 10, with a higher score meaning that the cancer tissue is more likely to spread.
Time Frame: Month 12
Population: Full Analysis Set included all participants with prostate cancer who signed informed consent and were randomised. Participants with missing Gleason score data are excluded.
Measure: Count of Participants; unit: Participants
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance
Number analyzed (Participants) | 26 | 34
Participants | 1 | 3

3. Secondary Outcome: Change From Baseline in the International Prostate Symptom Score (I-PSS) Total Symptom (S) Score
Description: The I-PSS is an 8-question tool used to measure prostate symptoms (≤7: mildly symptomatic; 8-19 moderately symptomatic; 20-35 severely symptomatic). The first 7 symptom questions answered on a scale of 0 (never) to 5 (almost always) are used to determine the I-PSS Total S Score for a total possible score of 0 to 35. The 8th question is quality of life and is not reported here. A negative change from baseline indicates improvement. An Analysis of Covariance (ANCOVA) model fitted with baseline I-PSS total score and age as covariates was used for analysis.
Time Frame: Baseline and Months 3, 6, 9 and 12
Population: Full Analysis Set included all participants with prostate cancer who signed informed consent and were randomised.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance
Number analyzed (Participants) | 58 | 57
score on a scale
  Change at Month 3 | 0.37 [-0.70 to 1.43] | 1.03 [-0.05 to 2.11]
  Change at Month 6 | -0.38 [-1.27 to 0.51] | 0.32 [-0.59 to 1.24]
  Change at Month 9 | -1.13 [-1.97 to -0.28] | 0.64 [-0.23 to 1.52]
  Change at Month 12 | -0.48 [-1.52 to 0.56] | 0.93 [-0.14 to 2.01]

4. Secondary Outcome: Prostatic Volume as a Measure of Tumor Radiologic Progression Using Dynamic Magnetic Resonance Imaging (MRI)
Description: MRI is an imaging technique used to investigate the anatomy and function of the body. Measurements were taken to calculate the prostatic volume in cubic millimeters (mm^3).
Time Frame: Baseline and Month 12
Population: Full Analysis Set included all participants with prostate cancer who signed informed consent and were randomised. Participants with missing MRI data are excluded from analyses. Number analyzed is the number of participants with prostatic volume data at the given time-point.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance
Number analyzed (Participants) | 56 | 57
mm^3
  Baseline: number analyzed (Participants) | 54 | 55
  Baseline | 48.48 (25.09) | 49.44 (25.88)
  Month 12: number analyzed (Participants) | 52 | 49
  Month 12 | 51.47 (28.15) | 48.33 (20.18)

5. Secondary Outcome: Highest Diameter of the Lesion as a Measure of Tumor Radiologic Progression Using Dynamic MRI
Description: MRI is an imaging technique used to investigate the anatomy and function of the body. Measurements were taken to determine the diameter of the lesions in millimeters (mm).
Time Frame: Baseline and Month 12
Population: Full Analysis Set included all participants with prostate cancer who signed informed consent and were randomized and for whom MRI was performed. Participants with missing MRI data are excluded from analyses. Number analyzed is the number of participants with diameter data at the given time-point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance
Number analyzed (Participants) | 56 | 57
mm
  Baseline: number analyzed (Participants) | 29 | 18
  Baseline | 6.39 (2.80) | 7.78 (2.02)
  Month 12: number analyzed (Participants) | 23 | 28
  Month 12 | 6.25 (3.62) | 7.69 (2.56)

6. Secondary Outcome: Change From Baseline in Prostate-specific Antigen (PSA) Levels
Description: Blood was collected and sent to a central laboratory for analysis of PSA reported in milligrams/milliliter (mg/mL). A negative change from baseline indicates improvement. An ANCOVA model fitted with baseline PSA Level and age as covariates was used for analyses.
Time Frame: Baseline and Months 3, 6, 9 and 12
Population: Full Analysis Set included all participants with prostate cancer who signed informed consent and were randomised.
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/mL
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance
Number analyzed (Participants) | 58 | 57
mg/mL
  Change at Month 3 | -4.61 [-5.07 to -4.15] | 0.22 [-0.25 to 0.70]
  Change at Month 6 | -3.27 [-3.95 to -2.59] | 0.85 [0.15 to 1.55]
  Change at Month 9 | -1.46 [-1.96 to -0.95] | 0.71 [0.20 to 1.21]
  Change at Month 12 | 0.17 [-0.69 to 1.04] | 0.76 [-0.13 to 1.66]

7. Secondary Outcome: Change From Baseline in Hospital Anxiety and Depression Scale (HADS) Score
Description: The HADS is a 14-item scale that measures anxiety (7-items) and depression (7-items) over the previous week. Each question is answered on a scale of 0 (best) to 3 (worst) for a total possible score of 0 to 42, with higher scores indicating more anxiety and depression. A negative change from baseline indicates improvement. An ANCOVA model fitted with baseline HADS score and age as covariates was used for analyses.
Time Frame: Baseline and Months 3, 6, 9 and 12
Population: Full Analysis Set included all participants with prostate cancer who signed informed consent and were randomised.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance
Number analyzed (Participants) | 58 | 57
score on a scale
  Change at Month 3 | -0.83 [-1.76 to 0.11] | -1.20 [-2.17 to -0.24]
  Change at Month 6 | -1.44 [-2.53 to -0.35] | -1.58 [-2.69 to -0.47]
  Change at Month 9 | -2.06 [-3.21 to -0.91] | -1.76 [-2.95 to -0.56]
  Change at Month 12 | -1.87 [-2.98 to -0.76] | -1.95 [-3.09 to -0.80]

8. Secondary Outcome: Change From Baseline in the International Index of Erectile Function (IIEF-5) Questionnaire Score
Description: The IIEF-5, a 5 question patient completed questionnaire, is a measure of erectile dysfunction over the past 6 months. Each question is answered on a scale of 1 (worst) to 5 (best). Total score ranges from 5 to 25 with higher scores indicating better function (5-7: severe; 8-11: moderate; 12-16: mild to moderate;17-21: mild; 22-25: none). A positive change from baseline indicates improvement. A negative change from baseline indicates a worsening. An ANCOVA model fitted with baseline IIEF-5 score and age as covariates was used for analyses.
Time Frame: Baseline and Months 3, 6, 9 and 12
Population: Full Analysis Set included all participants with prostate cancer who signed informed consent and were randomised.
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance
Number analyzed (Participants) | 58 | 57
score on a scale
  Change at Month 3 | -7.40 [-9.02 to -5.78] | 0.00 [-1.65 to 1.65]
  Change at Month 6 | -5.87 [-7.52 to -4.22] | 0.01 [-1.69 to 1.71]
  Change at Month 9 | -1.94 [-3.20 to -0.67] | -0.38 [-1.69 to 0.94]
  Change at Month 12 | -1.68 [-3.11 to -0.24] | -0.02 [-1.49 to 1.46]

ADVERSE EVENTS:
Time Frame: First dose of study drug to the End of Study Visit (Up to 12 Months)
Description: At each visit the investigator documented any occurrence of adverse events and abnormal laboratory findings. Any event reported by the participant or observed by the investigator was recorded.
Arm/Group | Leuprorelin 11.25 mg | Active Surveillance
Serious Adverse Events (participants affected / at risk) | 4/58 | 3/57
Other Adverse Events (participants affected / at risk) | 40/58 | 11/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin 11.25 mg (N=58) | Active Surveillance (N=57)
Atrial flutter (Cardiac disorders) | 1 | 0
Fatigue (Vascular disorders) | 1 | 0
Dizziness (Vascular disorders) | 1 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0
Erysipelas (Infections and infestations) | 0 | 1
Urinary tract disorder (Renal and urinary disorders) | 0 | 1
Pancreatic neoplasm (Gastrointestinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Leuprorelin 11.25 mg (N=58) | Active Surveillance (N=57)
Fatigue (General disorders) | 4 | 0
Bronchitis (Infections and infestations) | 3 | 2
Headache (Nervous system disorders) | 3 | 0
Erectile dysfunction (Psychiatric disorders) | 7 | 2
Dysuria (Renal and urinary disorders) | 4 | 2
Erectile dysfunction (Reproductive system and breast disorders) | 3 | 0
Hot flush (Reproductive system and breast disorders) | 17 | 0
Libido decreased (Reproductive system and breast disorders) | 6 | 0
Hot flush (Vascular disorders) | 6 | 0
Flushing (Vascular disorders) | 9 | 0
Hypertension (Vascular disorders) | 1 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.